CLINICAL TRIAL: NCT06409819
Title: Phase 1/ 2 Trial of Phage Therapy for Recurrent UTIs in Kidney Transplant Recipients
Brief Title: Phage Therapy for Recurrent UTIs in Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Saima Aslam, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 809673
Record Dates: First submitted 2024-04-23; First posted 2024-05-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Urinary Tract Infection, Recurrent
MeSH Terms: conditions — Urinary Tract Infections | interventions — Phage Therapy

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to phage therapy or placebo in a 2:1 fashion. Participants will be blinded to study assignment.
Who Masked: Participant
Masking Description: Both the phage preparation and placebo will be packaged as 1 ml clear solution in a plastic syringe. For safety, the pharmacy and research team will be aware of the assigned intervention. Only the participants will be blinded to study arm assignment. The effectiveness of the blinding process will be assessed by querying participants which intervention they think they received after the final participant has completed the 180-day study period by assessing the level of agreement between self-report and actual assignment.
  Study intervention will only be initiated while the participant is asymptomatic and does not have an active symptomatic UTI. Eligible participants will be randomized to phage therapy or placebo in a 2:1 fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention phage therapy (Active Comparator): Clear 1 milliliter (ml) solution in a plastic needless syringe. Phage therapy will consist of twice daily intravenous (IV) dose of previously selected phage combination of at least 109 plaque forming units (PFU)/ ml concentration per phage but not to exceed 5EU/Kg/hr of total lipopolysaccharide endotoxin for the entire dose as per FDA guidelines.
  Interventions: Drug: phage therapy
- Intervention control arm (normal saline placebo) (Placebo Comparator): Clear 1mL solution in a plastic needless syringe. Placebo will consist of IV normal saline administered in the same manner as the active comparator for 7 days.
  Interventions: Drug: control

INTERVENTIONS:
Drug: phage therapy — phage therapy will consist of a combination of three lytic phages that are active against the participant's E. coli isolates and will be administered intravenously twice daily for 7 days.
  Other Names: targeted phage therapy
  Arms: Intervention phage therapy
Drug: control — Participants assigned to the control arm will start a 7-day course of intravenous sterile normal saline (placebo) administered twice daily.
  Other Names: placebo
  Arms: Intervention control arm (normal saline placebo)

SUMMARY:
This proposal will take an important first step in the study of phage therapy for treatment of recurrent urinary tract infection (rUTI) in female kidney transplant recipients (KTR); a common condition that is associated with increasing multidrug resistance, sickness, loss of kidney function and death. The investigators will conduct a randomized phase I/II pilot clinical trial of targeted phage therapy versus placebo in asymptomatic female KTR with a history of rUTI due to Escherichia coli to assess safety, tolerability, and feasibility of this approach, possible efficacy, and changes in the gut and urinary microbiome during the 180 days of the study. This highly innovative and impactful proposal will provide proof of concept data and also inform the design of a subsequent larger phase III clinical trial of phage therapy for rUTI treatment in KTR and will have broad downstream effects within the fields of infectious diseases and transplantation.

DETAILED DESCRIPTION:
The overarching hypothesis is that phage therapy directed against E. coli in female KTR is safe and associated with a reduction in UTI event rate via a targeted impact on the gut and urinary microbiome. This is a Phase 1/ 2 randomized, placebo-controlled clinical trial.

* A description of methods to be used to minimize bias Participants will be randomized to one of 2 arms - one active intervention phage therapy and the second is active intervention control arm (normal saline placebo). Participants will not be aware of study assignment and the medication delivered to them will look identical - clear 1mL solution in a plastic needless syringe.
* The number of study groups/arms and study intervention duration:

  * Investigators plan to enroll participants that fulfill eligibility criteria until they reach their goal of 16 participants in each arm (total N= 32).

This clinical trial will evaluate the effect of phage only (without concomitant antibiotics) compared to placebo for UTI prevention in asymptomatic female KTR with a history of rUTI. There are no rigorous, published trials testing this approach, nor are there new therapeutics for rUTI in KTR on-market at this time. Most IND cases or trials compare phage plus antibiotic which limits the ability to isolate the contribution from phage to treatment success. The proposed research will utilize a phase I/II pilot trial designed to assess the safety, tolerability, and feasibility of therapy, compare potential efficacy, and assess changes to microbiome profiles in the female participants who will receive either phage or placebo. As the participants will be treated when they are asymptomatic, no active control is needed and so Investigators will use normal saline placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Female kidney transplant recipients, aged 18 and older with a confirmed diagnosis of a history of recurring UTI with E. coli as their typical uropathogen.
2. Two urine culture proven UTIs in prior 6 months or three in prior 12 months due to E coli. UTI is defined as any change in symptoms from baseline urinary comfort (dysuria, hematuria, abdominal/flank pain, increased urinary frequency) or systemic signs of infection (fever, chills, systemic inflammatory reaction syndrome etc.) associated with a positive urine culture with bacterial growth of ≥104 colony forming units/mL).
3. Ability to self-administer study drug (or a family member that will do so) and willing to adhere to the phage therapy regimen.
4. For participants able to become pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 months after the end of phage therapy administration.
5. Provision of signed and dated informed consent form
6. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Presents with hardware in the urinary tract (e.g. stent, percutaneous nephrostomy, chronic urinary catheter).
2. Recipient of >1 kidney transplant.
3. Recipient of Ileal conduit.
4. Recipient of surgical neobladder.
5. Diagnosed with chronic urinary retention requiring self-catheterization.
6. Anatomic cause for rUTI such as ureteral stenosis.
7. Within the first 3 months of kidney transplant.
8. Venous access sites or in whom an existing venous access site needs to be preserved for future need (as per the participant's transplant nephrologist/ surgeon)
9. Diagnosed with active cytomegalovirus or BK virus infections.
10. Current pregnancy, actively trying to conceive, or lactating.
11. Known allergic reactions to phage products.
12. Prisoners or individuals without decisional capacity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult cis-gender female kidney transplant recipients (KTRs) aged >18 years
Enrollment: 32 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 180 days
  Safety of phage administration will be assessed by the incidence of adverse events (AE) as assessed by CTCAE v4.0. As this is a phase 1/ 2 pilot clinical study, the primary outcome is safety and tolerability of the IP.
Enrollment Feasibility | 180 days
  Enrollment feasibility of the trial protocol will be assessed by enrollment and randomization (goal is ≥75% of target N at year 1 of the award).
Proportion of participants with a phage match | 180 days
  Proportion of participants with a phage match will be assessed by the number of enrolled participants with a phage match (goal is ≥70%).
Study Drug Adherence | 180 days
  Adherence to study drug administration by the participants (goal is ≥90%),

SECONDARY OUTCOMES:
Treatment Efficacy | 180 days
  Efficacy of the treatment as measured by the number of UTI events due to the original infecting pathogen over the 180-day study observation period (event rate), calculated for the intent to treat population. As this is a phase 1/ 2 trial, this outcome will give us an efficacy signal.
Desirability of Outcome Rankings (DOOR) Score | 180 days
  A graded outcome based on clinical and microbiological parameters
Proportion of Participants with UTI | 180 days
  The proportion of participants with UTI will be assessed.
Days to first symptomatic UTI from the original infecting pathogen | 180 days
  The number of days to first symptomatic UTI from the original infecting pathogen will be assessed.
Microbiological Eradication of Asymptomatic Bacteriuria | 180 days
  The microbiological eradication of asymptomatic bacteriuria will be assessed.
Need for intravenous (IV) antibiotics | 180 days
  The need for IV antibiotics will be assessed.
Number of days on antibiotics | 180 days
  The number of days on antibiotics will be assessed.
Emergency room visit/ hospitalization due to UTI | 180 days
  Any occurrence of emergency room visit/ hospitalization due to UTI will be assessed.
Change in kidney function from baseline to end of the study period | 180 days
  The change in kidney function from baseline to end of the study period will be assessed via serum creatinine, glomerular filtration rate, and occurrence of acute kidney injury.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States